CLINICAL TRIAL: NCT07129668
Title: Effects of Finger Kazoo Exercise With and Without Oropharyngeal Enlargement in the Operatic Singing Voice: A Randomized, Single-Blind, Crossover Controlled Clinical Trial
Brief Title: Effects of Finger Kazoo Exercise With and Without Oropharyngeal Enlargement in the Operatic Singing Voice
Acronym: FIKVOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: School of Health Sciences, University of Aveiro (ESSUA) (Unknown)
Responsible Party: Principal Investigator, Jean Carlos Gorges, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-CE/2025; doi.org/10.54499/2023.0361.BD (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Voice Alteration
Keywords: Singing Voice; Finger Kazoo; SOVTE; Operatic Voice
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: Fifteen classically trained singers participated in a randomized, single-blind, crossover trial with two experimental sessions separated by 48 hours. Participants were allocated via Sealed Envelope randomization to start in Condition A (without oropharyngeal expansion) or Condition B (with oropharyngeal expansion). In each session, standardised recordings were obtained before and after the intervention, including maximum phonation time for the vowels /a/ and /i/, and an operatic aria excerpt.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition A (Active Comparator): Without Oropharyngeal Enlargement
  Interventions: Behavioral: Condition A; Behavioral: Condition B
- Condition B (Active Comparator): With Oropharyngeal Enlargement
  Interventions: Behavioral: Condition A; Behavioral: Condition B
- Condition 0 or Baseline (Active Comparator): Condition 0 (Baseline) consists of producing the target vocal tasks without any semi-occlusion or intentional oropharyngeal modification just a pre vocal warmup.
  Interventions: Behavioral: Condition A; Behavioral: Condition B

INTERVENTIONS:
Behavioral: Condition A — Condition A consists of performing the Finger Kazoo exercise without inducing oropharyngeal enlargement. In this condition, participants place the index finger vertically in front of the lips to partially occlude the vocal tract, producing a semi-occluded vocal tract configuration, but without modifying tongue position, soft palate height, or pharyngeal wall expansion to increase the oropharyngeal space.
  Other Names: Whitout Oropharyngeal Enlargement
Behavioral: Condition B — Condition B consists of performing the Finger Kazoo exercise with intentional oropharyngeal enlargement. In this condition, participants place the index finger vertically in front of the lips to partially occlude the vocal tract, producing a semi-occluded vocal tract configuration, while simultaneously modifying tongue position, elevating the soft palate, and expanding the pharyngeal walls to increase the oropharyngeal space.
  Other Names: With Oropharyngeal Enlargement

SUMMARY:
This clinical trial aimed to evaluate the effects of the semi-occluded vocal tract exercise Finger Kazoo (FK), with and without oropharyngeal expansion, on the singing voice. Fifteen classically trained singers, screened using the Singing Voice Handicap Index-10 (SVHI-10), participated in a randomized, single-blind, crossover trial with two experimental sessions separated by 48 hours. Participants were randomized via Sealed Envelope to start in Condition A (without oropharyngeal expansion) or Condition B (with oropharyngeal expansion). In each session, standardized recordings were obtained before and after the intervention, including maximum phonation time for the vowels /a/ and /i/, and an operatic aria excerpt. Acoustic analysis (PRAAT) extracted fundamental frequency (F0), jitter, and shimmer. Comparisons between baseline and experimental conditions were performed using paired-samples t-tests, Wilcoxon tests, robust paired t-tests, and Friedman ANOVA with Durbin-Conover, Tukey, Bonferroni, and Holm post hoc corrections, with a 95% confidence interval. Auditory-perceptual evaluation was conducted by 15 blinded experts using the EAI Scale Form, with balanced sample distribution among raters. Self-perceptual evaluation was also performed by participants using the same scale.

ELIGIBILITY:
Inclusion Criteria:

* Classically trained singers aged 18 to 45 years.
* Scoring below the cutoff for vocal handicap on the Singing Voice Handicap Index-10 (SVHI-10 ≤ 6 )*.
* No history of recently vocal fold pathology or laryngeal surgery.
* Non-smokers and no current upper respiratory infection.
* Willingness and ability to attend two experimental sessions spaced 48 hours apart.

Exclusion Criteria:

* Presence of any current voice disorder or history of chronic laryngeal disease.
* Recent respiratory infection within 2 weeks prior to enrollment.
* Use of medications affecting voice or respiratory function.
* Inability or unwillingness to comply with study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-26 (Actual)

PRIMARY OUTCOMES:
Maximum Phonation Time (MPT) variation between conditions without and with oropharyngeal enlargement. | Baseline and 48 hours after first session (allowing return to baseline before second session).
  Assessment of the difference in maximum phonation time (in seconds) between two experimental conditions: without oropharyngeal enlargement (Condition A) and with oropharyngeal enlargement (Condition B), during sustained vowel phonation.
  Data Collection Method: Acoustic recordings obtained using Praat software. The MPT was measured from the onset of phonation to cessation, with participants instructed to sustain the vowel at comfortable pitch and loudness.
  Analysis Method: Robust Paired Samples T-Test comparing MPT between Condition A and Condition B. Effect sizes calculated using Cohen's d. Results Summary: Mean MPT was significantly higher in Condition B (+7.9 s; p < .001; d = 0.46), indicating improved phonatory efficiency.

SECONDARY OUTCOMES:
Change in Fundamental Frequency Stability (ΔF0) between conditions without and with oropharyngeal enlargement. | Baseline and 48 hours after first session (allowing return to baseline before second session).
  Evaluation of the mean variation in fundamental frequency (in Hz) from onset to end of sustained vowel phonation, comparing Condition A and Condition B.
  Data Collection Method: Praat software pitch analysis, extracting F0 mean values for initial and final 3 seconds of the sustained vowel, then calculating the difference (ΔF0).
  Analysis Method: Robust Paired Samples T-Test. Results Summary: ΔF0 was significantly lower in Condition B (-7.6 Hz; p < .001; d = 0.39), indicating greater pitch stability.

OTHER OUTCOMES:
Change in Jitter between conditions without and with oropharyngeal enlargement. | Baseline and 48 hours after first session (allowing return to baseline before second session).
  Percentage variation in jitter between the initial and final segments of sustained vowel phonation.
  Data Collection Method: Jitter (%) extracted from Praat software and compared between initial and final segments. ΔJitter calculated as final - initial.
  Analysis Method: Robust Paired Samples T-Test. Results Summary: ΔJitter was significantly reduced in Condition B (-1.3%; p < .001; d = 0.54), indicating improved micro-frequency stability.
Change in Shimmer between conditions without and with oropharyngeal enlargement. | Baseline and 48 hours after first session (allowing return to baseline before second session).
  Percentage variation in shimmer between the initial and final segments of sustained vowel phonation.
  Data Collection Method: Shimmer (%) extracted from Praat software and compared between initial and final segments. ΔShimmer calculated as final - initial.
  Analysis Method: Robust Paired Samples T-Test. Results Summary: ΔShimmer was significantly reduced in Condition B (-2.1%; p < .001; d = 0.57), suggesting improved amplitude stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Essua - University of Aveiro, Aveiro, Aveiro District, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional and legal restrictions on data privacy and protection as per the data protection agreement signed with the University of Aveiro.